CLINICAL TRIAL: NCT00572468
Title: Pre-Operative Statin Therapy Versus Placebo in Human Prostate Cancer
Brief Title: Statin Therapy Versus Placebo Prior to Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CLIN-013-07S; VA IRB#1735 (Other: VA IRB); SOL-07130-L (Other: OHSU Knight Cancer Institute Identifier)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Cancer; Prostate Cancer
Keywords: cancer; pre-operative surgery; prostate; prostatectomy; radiation
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): Twenty-two men will be on the Statin arm and take 40 mg of simvastatin.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Twenty-two men will be on the placebo arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40 mg of simvastatin
  Other Names: statin
  Arms: Simvastatin
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
This is a randomized trial comparing the effect of oral simvastatin versus placebo on targets of the mevalonate pathway in men undergoing a prostatectomy as planned management for prostate cancer. Observed tissue effects will be correlated with changes in serum cholesterol and low-density lipoprotein.

DETAILED DESCRIPTION:
Prostate cancer patients that have chosen to undergo a prostatectomy as their primary treatment option will be recruited to this trial. Forty-four subjects will be randomized to either placebo or simvastatin (40 mg po/day) for 4 weeks prior to surgery. Serum samples will be obtained at baseline and immediately prior to prostatectomy. At prostatectomy, cancerous and benign prostate tissue will be microdissected and cryopreserved. Archival prostatectomy tissues will be used to construct tissue microarrays containing matched benign and malignant sections. The effect of HMG-CoA reductase inhibition on lipid raft cholesterol content and targets of prenylation will be determined. The incidence of apoptosis will be determined along with protein levels of mediators of apoptosis. Lastly the effect of statin therapy on cellular markers of proliferation will be determined.

Previously, we studied the effect of statin use on the risk of prostate cancer detection in a case-control study at the Portland VA Medical Center. Statin use was associated with a 62% reduction in cancer odds-risk (OR = 0.38, 95% CI 0.21-0.69). Although these epidemiologic and laboratory findings have generated enthusiasm for the study of statins in prostate cancer, no studies have examined the biologic effects of statins on prostate cancer in humans.

Hypothesis: Statin therapy prior to prostatectomy will successfully target the mevalonate pathway in the human prostate and this intervention will favorably alter tumor biomarker status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostatic adenocarcinoma with Gleason 5 to 7 (3+4 = 7 accepted, not 4 + 3 = 7)
* Radical prostatectomy chosen as primary treatment for prostate cancer
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Other preoperative or prior treatment directed at prostate cancer (i.e., Radiation, hormonal therapy, cryotherapy)
* Significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* History of or active liver disease or abnormal results of the baseline liver function test (> 2 x normal)
* Current use of:

  * simvastatin
  * lovastatin
  * other HMG-CoA inhibitors
  * lipid-lowering agents
  * Amiodarone
  * Cholestyramine
  * Cholestyramine and colestipol (bile acid sequestrants)
  * Clofibrate and fenofibrate
  * Cyclosporine
  * CYP3A4 inhibitors
  * Danazol
  * Diltiazem
  * Gemfibrozil
  * Niacin ( 1 g/day)
  * Verapamil and Warfarin
* Known allergy or sensitivity to ingredients in simvastatin

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-12; Primary Completion 2013-04 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Garzotto, MD, Principal Investigator — VA Medical Center, Portland
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Medical Center, Portland, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin: Participants were randomized into the Simvastatin arm of this trial.
- Placebo: Participants were randomized into the placebo arm of this trial.
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 22 | 20
Completed | 20 | 16
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: Years] | 60.4 [46 to 71] | 60.75 [53 to 73] | 60.56 [46 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 16 | 36
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Measure the Effect of Pre-operative Simvastatin Versus Placebo on the Mevalonate Pathway Synthesis and Target Activation in Benign and Malignant Prostate Tissue.
Description: Measure the effect of pre-operative simvastatin versus placebo on the mevalonate pathway synthesis and target activation in benign and malignant prostate tissue using Androgen Receptor (AR) antibody. AR was measured in tissue obtained at the time of prostatectomy in both benign and malignant tissues.
Time Frame: 5 years
Population: We enrolled a total of 42 subjects, 36 completed this study. Of the 36 subjects who completed this study, only 26 subjects had tissue available for this analysis.
Measure: Mean (95% Confidence Interval); unit: Percentage of cells
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 15 | 11
Percentage of cells | 168.6666667 [142.4517 to 194.882] | 182.7272727 [161.46353 to 203.99107]

2. Secondary Outcome: Compare the Effect of Pre-operative Simvastatin Versus Placebo on Prostate Cancer Cell Apoptosis and Its Mediators in Men Undergoing Planned Prostatectomy.
Description: Compare the effect of pre-operative simvastatin versus placebo on prostate cancer cell apoptosis and its mediators in men undergoing planned prostatectomy. Apoptosis was measured by calculating the percent of Ki67 cellular staining.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of cells
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 15 | 11
Percentage of cells | 7.53333 [3.95134 to 11.11532] | 6 [1.87843 to 10.12157]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline, weekly while on treatment, and at 30-day follow-up. Subjects were on trial for 4-8 weeks (depending on prostatectomy scheduling).
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 11/20 | 3/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=20) | Placebo (N=16)
UTI (Renal and urinary disorders) | 4 (4) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter discomfort (Renal and urinary disorders) | 1 (1) | 1 (1)
Bloody drainage from wound (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No